CLINICAL TRIAL: NCT06963710
Title: A Randomized, Double-Blind, Active-Controlled Multicenter Phase 2 Study Evaluating the Efficacy and Safety of ALG-000184 Compared With Tenofovir Disoproxil Fumarate in Untreated HBeAg-Positive and HBeAg-Negative Adult Subjects With Chronic Hepatitis B Virus Infection (B-SUPREME)
Brief Title: A Study Evaluating the Efficacy and Safety of ALG-000184 Compared With Tenofovir Disoproxil Fumarate in Untreated HBeAg-Positive and HBeAg- Negative Adult Subjects With Chronic Hepatitis B (B-SUPREME)
Acronym: B-SUPREME
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aligos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALG-000184-202
Record Dates: First submitted 2025-04-22; First posted 2025-05-09 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-04

CONDITIONS: Chronic Hepatitis B Infection
Keywords: Capsid Assembly Modulators; CAMs; CHB; HBV; Chronic Hepatitis B; Hepatitis B Infection; Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALG-000184 (Experimental): Orally for 48 weeks followed by open-label treatment with ALG-000184 for 48 weeks.
  Interventions: Drug: ALG-000184
- TDF (Active Comparator): Orally for 48 weeks followed by open-label treatment with ALG-000184 for 48 weeks.
  Interventions: Drug: TDF

INTERVENTIONS:
Drug: ALG-000184 — 300 mg tablet
  Arms: ALG-000184
Drug: TDF — 300 mg tablet
  Arms: TDF

SUMMARY:
This is a Phase 2 study to evaluate efficacy and safety of 48 weeks of oral once daily monotherapy with ALG-000184 versus tenofovir disproxil fumarate (TDF) for chronic HBV infection.

DETAILED DESCRIPTION:
This is a randomized, double-blind, active-controlled, multicenter Phase 2 study to evaluate the efficacy and safety of 48 weeks of oral (PO) once daily (QD) monotherapy with ALG-000184 versus TDF in treatment naive (TN) or currently not treated (CNT) HBeAg-positive and HBeAg-negative subjects with chronic HBV infection (inclusive of chronic infection and/or chronic hepatitis).

A total of approximately 200 eligible subjects will be enrolled across 2 study parts. Part 1 will be an evaluation of HBeAg-positive subjects with chronic HBV infection and Part 2 will be an evaluation of HBeAg-negative subjects with chronic HBV infection. Each study part will consist of a main study and an exploratory liver biopsy sub-study.

Following the 48-week double-blind dosing period (Week 48), all participating subjects (in Parts 1 and 2) will be allowed to roll over into a 48 week (i.e., Week 48-96) open-label treatment extension period where they will all receive ALG-000184 monotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female between 18 and 65 years of age, with body mass index (BMI) of 18.0 to 35.0 kg/m2 (or minimun age by local regulatory requirements).
2. HBeAg-positive and anti-HBeAg (HBeAb) negative (Part 1); or HBeAg-negative (Part 2).
3. HBsAg ≥LLOQ.
4. HBV DNA ≥20,000 IU/mL.
5. A history of a clinical diagnosis of chronic HBV infection AND an ALT values of ≤8×ULN during screening.
6. Must have the following chronic hepatitis B virus infection treatment status at screening:

   1. Have never received treatment with HBV antiviral medicines (NA, interferon) or investigational anti-HBV agents including a CAM [i.e., Treatment Naïve (TN) subjects], OR
   2. Have not been on treatment with approved (NA, interferon) or investigational HBV antiviral medicines (e.g., antisense oligonucleotides or small interfering RNAs) within 6 months or 5 half-lives (whichever is longer) prior to randomization (i.e., Currently Not Treated (CNT) subjects).

Key Exclusion Criteria:

1. Co-infection with hepatitis A, C, D, E or HIV or any evidence of clinically significant liver disease of non-HBV etiology.
2. Positive for anti-HBs antibodies.
3. History or current evidence of cirrhosis.
4. Liver fibrosis that is classified as Metavir Score ≥F3 liver disease.
5. History of, or current evidence of, hepatic decompensation.
6. Evidence of hepatocellular carcinoma (HCC) on a liver ultrasound.
7. Having received an investigational medicinal product or device within 4 weeks (or 5 half-lives, whichever is longer) before the planned first dose of study drug
8. Exclusionary screening laboratory values include:

   1. Aspartate aminotransferase (AST) >8×ULN,
   2. Bilirubin (total, direct) >1.2×ULN (unless Gilbert's syndrome is suspected)
   3. International Normalization Ratio (INR) >1.2×ULN

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
HBeAg positive: HBV DNA <Lower Limit of Quantification [LLOQ] (10 IU/mL, target detected or target not detected) | 48 weeks
  HBV DNA <Lower Limit of Quantification [LLOQ] (10 IU/mL, target detected or target not detected) at Week 48
HBeAg negative: HBV DNA <Lower Limit of Quantification [LLOQ] (10 IU/mL, target not detected) | 48 weeks
  HBV DNA <Lower Limit of Quantification [LLOQ] (10 IU/mL, target not detected) at Week 48

SECONDARY OUTCOMES:
Safety and Tolerability | 96 Weeks
  Number of participants with Treatment Emergent Adverse Events (TEAEs), with abnormal 12-lead electrocardiogram readings and abnormal clinical laboratory results.
HBV DNA levels | 48 weeks
  Categorized by HBV DNA ≥ Lower Limit of Quantification [LLOQ], HBV DNA <Lower Limit of Quantification [LLOQ] (target detected), and HBV DNA < Lower Limit of Quantification [LLOQ] (target not detected)
HBV DNA < lower limit of quantification [LLOQ] (target detected or target not detected) [HBeAg positive] | 48 weeks
  HBV DNA < Lower Limit of Quantification [LLOQ] (target detected or target not detected) at various time points during the first 48 weeks
HBV DNA < Lower Limit of Quantification [LLOQ] (target not detected) [HBeAg negative] | 48 weeks
  HBV DNA < Lower Limit of Quantification [LLOQ] (target not detected) at various time points during the first 48 weeks
Change in HBV DNA levels from baseline | 48 weeks
  Change from baseline in HBV DNA at various time points during the first 48 weeks.
Time to HBV DNA level <Lower Limit of Quantification [LLOQ] | 96 Weeks
  Time to HBV DNA < Lower Limit of Quantification [LLOQ] (target detected or target not detected) (HBeAg positive) and HBV DNA < Lower Limit of Quantification [LLOQ] (target not detected) (HBeAg negative)
Change in HBV RNA levels from baseline | 48 weeks
  Change from baseline in HBV RNA levels at various time points during the first 48 weeks
Time to HBV RNA level <Lower Limit of Quantification [LLOQ] | 96 Weeks
  Time to HBV RNA < Lower Limit of Quantification [LLOQ]
Subjects with abnormal ALT at baseline who have normal ALT at Week 48 | 48 weeks
  Subjects with abnormal ALT at baseline who have normal ALT at Week 48
Emergence of treatment associated mutations in the HBV genome | 96 Weeks
  Emergence of treatment associated mutations in the HBV genome
PK parameters of ALG-001075 | 96 Weeks
  PK parameters of ALG-001075 including the trough plasma concentration (Ctrough)
PK parameters of ALG-001075 | 96 Weeks
  PK parameters of ALG-001075 including the time to reach the maximum plasma concentration (Tmax)
PK parameters of ALG-001075 | 96 Weeks
  PK parameters of ALG-001075 including the maximum drug concentration (Cmax)
PK parameters of ALG-001075 | 96 Weeks
  PK parameters of ALG-001075 including the minimum drug concentration (Cmin)
PK parameters of ALG-001075 | 96 Weeks
  PK parameters of ALG-001075 including the area under the plasma concentration-time curve steady state (AUCss)
PK parameters of ALG-001075 | 96 Weeks
  PK parameters of ALG-001075 including the half-life

OTHER OUTCOMES:
Change in levels of various HBV antigens at various time points from Baseline | 96 Weeks
  Change from baseline in levels of various HBV antigens
Histologic, virologic, immunologic and/or PK-related endpoints | 96 Weeks
  Change in intrahepatic viral markers (e.g., HBV nucleic acid and antigen levels), immune cell populations, and inflammation/fibrosis biomarkers

CONTACTS AND LOCATIONS:
Locations (56):
- United States (17):
  - Aligos Investigational Site, Chandler, Arizona
  - Aligos Investigational Site, Coronado, California
  - Aligos Investigational Site, Garden Grove, California
  - Aligos Investigational Site, Los Angeles, California
  - Aligos Investigational Site, Palo Alto, California
  - Aligos Investigational Site, Pasadena, California
  - Aligos Investigational Site, Rialto, California
  - Aligos Investigational Site, San Francisco, California
  - Aligos Investigational Site, San Jose, California
  - Aligos Investigational Site, Miami, Florida
  - Aligos Investigational Site, Marrero, Louisiana
  - Aligos Investigational Site, Baltimore, Maryland
  - Aligos Investigational Site, Chevy Chase, Maryland
  - Aligos Investigational Site, Boston, Massachusetts
  - Aligos Investigational Site, Manhasset, New York
  - Aligos Investigational Site, New York, New York
  - Aligos Investigational Site, Durham, North Carolina
- Bulgaria (3):
  - Aligos Investigational Site, Sliven
  - Aligos Investigational Sites, Sofia
  - Aligos Investigational Site, Stara Zagora
- Canada (4):
  - Aligos Investigational Site, Edmonton
  - Aligos Investigational Site, Ottawa
  - Aligos Investigational Site, Toronto
  - Aligos Investigational Sites, Vancouver
- China (6):
  - Aligos Investigational Sites, Beijing
  - Aligos Investigational Site, Chengdu
  - Aligos Investigational Site, Chongqing
  - Aligos Investigational Sites, Guangzhou
  - Aligos Investigational Site, Nanjing
  - Aligos Investigational Sites, Shanghai
- France (6):
  - Aligos Investigational Site, Clichy
  - Aligos Investigational Site, Limoges
  - Aligos Investigational Site, Nice
  - Aligos Investigational Site, Rennes
  - Aligos Investigational Site, Rouen
  - Aligos Investigational Site, Toulouse
- Aligos Investigational Sites, Hong Kong, Hong Kong
- Aligos Investigational Site, Milan, Italy
- Aligos Investigational Site, Chisinau, Moldova
- Aligos Investigational Site, Auckland, New Zealand
- Aligos Investigational Sites, Bucharest, Romania
- South Korea (5):
  - Aligos Investigational Site, Ansan
  - Aligos Investigational Site, Busan
  - Aligos Investigational Sites, Seoul
  - Aligos Investigational Site, Ulsan
  - Aligos Investigational Site, Yangsan
- Spain (2):
  - Aligos Investigational Site, Barcelona
  - Aligos Investigational Site, Pontevedra
- Taiwan (5):
  - Aligos Investigational Site, Chiayi City
  - Aligos Investigational Site, Kaohsiung City
  - Aligos Investigational Site, Taichung
  - Aligos Investigational Site, Tainan
  - Aligos Investigational Site, Taipei
- United Kingdom (3):
  - Aligos Investigational Site, Glasgow
  - Aligos Investigational Site, Leicester
  - Aligos Investigational Sites, London